CLINICAL TRIAL: NCT00689884
Title: A Prospective Feasibility and Cost Analysis of Peripheral Blood Stem Cell Mobilization Using Pegfilgrastim in Patients With Hematologic Malignancies
Brief Title: Feasibility and Cost Analysis of PBSC Mobilization Using Pegfilgrastim in Hematologic Malignancies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, John M. Hill, Jr., MD, Director, Allogeneic Bone Marrow Transplant Program, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0546
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group A (Experimental): All eligible patients will receive chemotherapy and one dose of Pegfilgrastim
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Pegfilgrastim — Pegfilgrastim: Sub Cutaneous, 6 mg on Day 3 of chemotherapy regimen or as otherwise indicated by chemotherapy regimen (ie., 24 hours after completion of chemotherapy).
  Other Names: Neulasta

SUMMARY:
The purpose of this study is to determine the efficacy of Pegfilgrastim in the mobilization of autologous peripheral blood stem cells (PBSCs), defined as cell yield ≥ 3 x 10e6 CD34+/kg and to assess the costs related to Pegfilgrastim use in the mobilization of autologous PBSCs. Also to determine the side effects of Pegfilgrastim in the mobilization of autologous peripheral blood stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with hematologic malignancies undergoing stem cell mobilization in association with chemotherapy, prior to autologous stem cell transplantation.
2. Prior Treatment:No parenteral cytotoxic chemotherapy within 2 weeks prior to initiation of chemo-mobilization therapy.
3. Performance Status: Karnofsky > 70%
4. Age >18
5. Life Expectancy > 4 months
6. Bone Marrow: bone marrow biopsy and aspirate
7. Blood counts: The patient must have adequate bone marrow function, i.e. a total WBC of > 2,000/ul, a Hgb of > 7 g/dl, and a platelet count of > 50,000/ul, unless this abnormality is believed to be due to the underlying disease.
8. Pulmonary function tests: DLCO > 55% predicted.
9. Cardiac: Left ventricular ejection fraction of > 40% by radionuclide scan or echocardiography.
10. Liver function tests (bilirubin, alkaline phosphatase, and SGOT/SGPT) < 3 x normal (unless believed to be elevated due to disease).
11. Renal function (24 hour urine for creatinine clearance, if clinically indicated): The patient must have adequate renal function (creatinine clearance >50 ml/min), except when renal insufficiency is felt related to the underlying malignancy.
12. No significant co-morbid medical or psychiatric illness that would significantly compromise the patient's clinical care and chances of survival in the transplant setting.
13. No significant established splenomegaly (i.e. spleen size > 20 cm)
14. Informed written consent must be obtained. Patients must be able to give informed consent as a prerequisite to this procedure. The Informed Consent form will become part of his/her permanent record and a copy will be given to the patient.

Exclusion Criteria:

1. Patients with greater than three pre-transplant chemotherapy regimens and/or poor stem cell reserve as demonstrated by significant marrow hypocellularity (<20%) will not be mobilized on the first phase regimen
2. Medical, social, or psychological factors that would prevent the patient from receiving or cooperating with the full course of therapy.
3. Evidence on physical exam, LP, CT, or MRI scan of CNS involvement with malignancy.
4. Uncontrolled or severe cardiovascular disease, including recent (< 6 months) myocardial infarction, congestive heart failure, angina (symptomatic despite optimal medical management), life-threatening dysrhythmia, or clinically significant obstructive/restrictive pulmonary disease.
5. Serology positive for HIV.
6. Positive pregnancy test or presence of lactation.
7. Uncontrolled active infection.
8. Documented hypersensitivity to any of the drugs used in the protocol.
9. No concomitant,ongoing malignancy that is life-threatening, based on PI's evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Hill Jr., MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy Plus Pegfilgrastim: All eligible patients will receive chemotherapy and one dose of Pegfilgrastim
Period: Overall Study
Arm/Group | Chemotherapy Plus Pegfilgrastim
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy Plus Pegfilgrastim
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Pegfilgrastim in the Mobilization of Autologous Peripheral Blood Stem Cells (PBSCs), Defined as Cell Yield ≥ 3 x 10e6 CD34+/kg
Description: Outcome was not reported. The study was terminated for lack of enrollment. Data collection was terminated. No data analysis was performed.
Time Frame: 2 years
Population: Outcome was not reported. The study was terminated for lack of enrollment. Data collection was terminated. No data analysis was performed.
Groups:
- Chemotherapy Plus Pegfilgrastim: Outcome was not reported. The study was terminated for lack of enrollment. Data collection was terminated. No data analysis was performed.
Arm/Group | Chemotherapy Plus Pegfilgrastim
Number analyzed (Participants) | 0

2. Secondary Outcome: Assess the Per-patient Costs Related to Pegfilgrastim Use in the Mobilization of Autologous PBSCs in 16 Study Participants.
Description: Costs will be divided into three categories: 1. Pre-pheresis preparation (cost of Pegfilgrastim, laboratory testing, drug administration, providers, line placement); 2. Pheresis procedure (costs related to # collections and total hours on apheresis machine, microbiological testing, provider, CD34 analysis and related labs, cryopreservation/storage and complications); 3. Post-pheresis processing (cost of stem cell thawing, microbiological testing, CD34 analysis and related labs, providers, administration).
Time Frame: At each stage of pheresis for each enrolled subject for a maximum of 2 years.
Population: as for outcome 1
Groups:
- Group 1: Outcome was not reported. The study was terminated for lack of enrollment. Data collection was terminated. No data analysis was performed.
Arm/Group | Group 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No adverse event data was collected
Arm/Group | Chemotherapy Plus Pegfilgrastim
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Outcome was not reported. The study was terminated for lack of enrollment. Data collection was terminated. No data analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No